CLINICAL TRIAL: NCT02853760
Title: Affective Responses in Mountain Hiking: A Randomized Controlled Trial Focusing on Differences Between Indoor and Outdoor Activity
Brief Title: Affective Responses in Mountain Hiking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Martin Burtscher, Prof, Universitaet Innsbruck
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ARMH
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Affect
MeSH Terms: interventions — Walking; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Outdoor mountain hiking (M) (Experimental): First part of the intervention: an uphill walking phase on single trails and forest roads in a sparse forest with view on the mountainous region around Innsbruck for 6 km in around 1.5 hours together with the test leader. Regarding the walking intensity, the participants were instructed to choose a "brisk without overspending" pace (average speed: 4 km/h).
  In the second part of the intervention, the participants were walking downhill on the same track for around 70 minutes back to the starting point to respond to the post-test (average speed: 5.2 km/h).
  Interventions: Behavioral: walking
- Indoor treadmill walking (T) (Active Comparator): To ensure that all physical parameters were simultaneous to the outdoor mountain hiking condition, the distance, the difference in height, the average inclination of the track, and the time needed for the outdoor mountain hiking situation were measured in a pilot study.
  First part: uphill walking, inclination: 10%, time: 1.5 hours, and speed: 4 km/h (resulting in 600 m difference in height). In accordance to possible differences in outdoor speed, the participants were allowed to change the treadmill's speed in a small range (3.8 to 4.2 km/h) to adapt to the wording "brisk without overspending". Second part of the intervention contained 70 minutes of level walking on the same treadmills (5.2 km/h, 6km).
  Interventions: Behavioral: walking; Device: Treadmill
- Sedentary control condition (C) (No Intervention): The sedentary control situation was located in a quiet room at the university with access to computers. The participants were allowed to use the computers, to read, and to talk, but had to remain in a sedentary position. To control for possible differences in affective response due to the daytime, the sedentary control condition contained the same timing of the measurements than the intervention condition. Sociodemographic data were collected for 5 to 10 minutes in this condition using a web-based questionnaire.

INTERVENTIONS:
Behavioral: walking
  Arms: Indoor treadmill walking (T); Outdoor mountain hiking (M)
Device: Treadmill
  Arms: Indoor treadmill walking (T)

SUMMARY:
Using a within-subject design, 42 healthy participants were randomly exposed to three different conditions: outdoor mountain hiking, indoor treadmill walking, and sedentary control situation (3.5 hours each). Measures included the Feeling Scale, Felt Arousal Scale and a Mood Survey Scale. Univariate ANOVAs were used to analyse differences between the conditions.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation

Exclusion Criteria:

* pregnancy
* breast-feeding
* chronic or acute diseases (already existing or diagnosed during the study)
* age below 18 and above 70 years
* unable to be physically active assessed by the Physical Activity Readiness Questionnaire (Shephard, Thomas, & Weller, 1991)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kopp, Prof., Study Director — martin.kopp@uibk.ac.at

REFERENCES:
- [Result] Niedermeier M, Einwanger J, Hartl A, Kopp M. Affective responses in mountain hiking-A randomized crossover trial focusing on differences between indoor and outdoor activity. PLoS One. 2017 May 16;12(5):e0177719. doi: 10.1371/journal.pone.0177719. eCollection 2017. PMID 28520774
- [Result] Niedermeier M, Grafetstatter C, Hartl A, Kopp M. A Randomized Crossover Trial on Acute Stress-Related Physiological Responses to Mountain Hiking. Int J Environ Res Public Health. 2017 Aug 11;14(8):905. doi: 10.3390/ijerph14080905. PMID 28800067

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As the project was a randomized crossover study, all participants were exposed to all three conditions.
Groups:
- Sequence Group MTC: All participants were exposed to three different conditions in a randomized starting order: outdoor mountain hiking (M), indoor treadmill walking (T), and sedentary control situation (C) (approximately three hours each).
  The order of conditions of the present group was M, followed by T, followed by C.
- Sequence Group MCT: All participants were exposed to three different conditions in a randomized starting order: outdoor mountain hiking (M), indoor treadmill walking (T), and sedentary control situation (C) (approximately three hours each).
  The order of conditions of the present group was M, followed by C followed by T.
- Sequence Group TMC: All participants were exposed to three different conditions in a randomized starting order: outdoor mountain hiking (M), indoor treadmill walking (T), and sedentary control situation (C) (approximately three hours each).
  The order of conditions of the present group was T, followed by M, followed by C.
- Sequence Group TCM: All participants were exposed to three different conditions in a randomized starting order: outdoor mountain hiking (M), indoor treadmill walking (T), and sedentary control situation (C) (approximately three hours each).
  The order of conditions of the present group was T, followed by C, followed by M.
- Sequence Group CTM: All participants were exposed to three different conditions in a randomized starting order: outdoor mountain hiking (M), indoor treadmill walking (T), and sedentary control situation (C) (approximately three hours each).
  The order of conditions of the present group was C, followed by T, followed by M.
- Sequence Group CMT: All participants were exposed to three different conditions in a randomized starting order: outdoor mountain hiking (M), indoor treadmill walking (T), and sedentary control situation (C) (approximately three hours each).
  The order of conditions of the present group was C, followed by M, followed by T.
Period: First Intervention (3 Hours)
Arm/Group | Sequence Group MTC | Sequence Group MCT | Sequence Group TMC | Sequence Group TCM | Sequence Group CTM | Sequence Group CMT
Started | 7 | 10 | 7 | 8 | 8 | 7
Completed | 7 | 10 | 7 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence Group MTC | Sequence Group MCT | Sequence Group TMC | Sequence Group TCM | Sequence Group CTM | Sequence Group CMT
Started | 7 | 10 | 7 | 8 | 8 | 7
Completed | 7 | 10 | 6 | 6 | 8 | 5
Not Completed | 0 | 0 | 1 | 2 | 0 | 2
Not completed — acute illness (not connected with the study) | 0 | 0 | 1 | 2 | 0 | 2
Period: Second Intervention (3 Hours)
Arm/Group | Sequence Group MTC | Sequence Group MCT | Sequence Group TMC | Sequence Group TCM | Sequence Group CTM | Sequence Group CMT
Started | 7 | 10 | 6 | 6 | 8 | 5
Completed | 7 | 10 | 6 | 6 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence Group MTC | Sequence Group MCT | Sequence Group TMC | Sequence Group TCM | Sequence Group CTM | Sequence Group CMT
Started | 7 | 10 | 6 | 6 | 8 | 5
Completed | 7 | 10 | 6 | 6 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (3 Hours)
Arm/Group | Sequence Group MTC | Sequence Group MCT | Sequence Group TMC | Sequence Group TCM | Sequence Group CTM | Sequence Group CMT
Started | 7 | 10 | 6 | 6 | 8 | 5
Completed | 7 | 10 | 6 | 6 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As the project was a randomized crossover study, all participants were exposed to all three conditions. The baseline data of all participants were combined in one Arm/Group ("All Study Participants").
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 42

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Subscales of Mood Survey Scale at 3 Hours
Description: Mood Survey Scale, min: 5, max: 25 higher score: better outcome All Outcome Measures are reported "per intervention", i.e., the data in Arms/Groups reflect the participants of the particular intervention.
Time Frame: baseline and 3 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Outdoor Mountain Hiking (M): First part of the intervention: an uphill walking phase on single trails and forest roads in a sparse forest with view on the mountainous region around Innsbruck for 6 km in around 1.5 hours together with the test leader. Regarding the walking intensity, the participants were instructed to choose a "brisk without overspending" pace (average speed: 4 km/h).
  In the second part of the intervention, the participants were walking downhill on the same track for around 70 minutes back to the starting point to respond to the post-test (average speed: 5.2 km/h).
  walking
- Indoor Treadmill Walking (T): To ensure that all physical parameters were simultaneous to the outdoor mountain hiking condition, the distance, the difference in height, the average inclination of the track, and the time needed for the outdoor mountain hiking situation were measured in a pilot study.
  First part: uphill walking, inclination: 10%, time: 1.5 hours, and speed: 4 km/h (resulting in 600 m difference in height). In accordance to possible differences in outdoor speed, the participants were allowed to change the treadmill's speed in a small range (3.8 to 4.2 km/h) to adapt to the wording "brisk without overspending". Second part of the intervention contained 70 minutes of level walking on the same treadmills (5.2 km/h, 6km).
  walking
  Treadmill
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
Number analyzed (Participants) | 42 | 42 | 42
score on a scale | 0.54 (3.73) | -1.27 (3.79) | -2.22 (3.84)

2. Primary Outcome: Change From Baseline Feeling Scale at 3 Hours
Description: Feeling Scale, min: -5, max: +5 higher score: better outcome All Outcome Measures are reported "per intervention", i.e., the data in Arms/Groups reflect the participants of the particular intervention.
Time Frame: baseline and 3 hours after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
Number analyzed (Participants) | 42 | 42 | 42
units on a scale | 1.37 (1.66) | 0.36 (2.07) | -0.81 (1.77)

3. Primary Outcome: Change From Baseline Felt Arousal Scale at 3 Hours
Description: Felt Arousal Scale, min: 0, max: 6 higher score: better outcome All Outcome Measures are reported "per intervention", i.e., the data in Arms/Groups reflect the participants of the particular intervention.
Time Frame: baseline and 3 hours after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
Number analyzed (Participants) | 42 | 42 | 42
units on a scale | 0.15 (1.45) | -0.19 (1.50) | -0.57 (1.06)

4. Secondary Outcome: Change From Baseline Blood Pressure at 3 Hours
Description: All Outcome Measures are reported "per intervention", i.e., the data in Arms/Groups reflect the participants of the particular intervention.
Time Frame: baseline and 3 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
Number analyzed (Participants) | 41 | 42 | 42
mmHg | -6.08 (10.16) | -4.53 (8.32) | -1.83 (9.81)

5. Secondary Outcome: Change From Baseline Heart Rate Variability at 3 Hours
Description: as for outcome 4
Time Frame: baseline and 3 hours
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
Number analyzed (Participants) | 41 | 42 | 41
ms | 10.16 (46.43) | 5.75 (31.14) | 15.06 (21.45)

6. Secondary Outcome: Change From Baseline Cortisol at 3 Hours (Saliva Sampling)
Description: as for outcome 4
Time Frame: baseline and 3 hours
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
Number analyzed (Participants) | 42 | 42 | 42
nmol/l | -2.98 (3.49) | -3.12 (3.41) | -2.00 (2.85)

ADVERSE EVENTS:
Time Frame: During the 3 interventions and the measurements, approximately 3.5 hours each. During the 2 washout phases, approximately 1 week each, by self-report of the participants.
Arm/Group | Outdoor Mountain Hiking (M) | Indoor Treadmill Walking (T) | Sedentary Control Condition (C)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42

LIMITATIONS AND CAVEATS:
* not feasible to apply downhill walking in the indoor situation, which resulted in a slightly different form of physical activity during the second part of the intervention
* affective responses might be influenced by at least two confounding variables: the level of social interaction and the intensity of PA.
* we did not include a follow-up measurement
* we are aware about a possible selection bias in the present study
* the length of the washout phase was not the same in all subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No